CLINICAL TRIAL: NCT05845658
Title: A Randomized, Double-Blind Sham Controlled Clinical Trial to Evaluate The Efficacy of Electrical Vestibular Stimulation (VeNS), Compared to a Sham Control For The Management Of Anxiety
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Treatment for Anxiety: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: R D Gardi Medical College, Ujjain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICNAS001
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VeNS (Active Comparator): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Active VeNS
- Sham VeNS (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Sham VeNS

INTERVENTIONS:
Device: Active VeNS — The VeNS device utilizes a technology called galvanic vestibular stimulation (GVS) (sometimes termed vestibular nerve stimulation (VeNS)). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Arms: Active VeNS
Device: Sham VeNS — The VeNS device utilizes a technology called galvanic vestibular stimulation (GVS) (sometimes termed vestibular nerve stimulation (VeNS)). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Arms: Sham VeNS

SUMMARY:
The present study will be conducted at the Department of Physiology in collaboration with the Department of Psychiatry of R.D. Gardi Medical College, Ujjain, Madhya Pradesh.

This double-blind randomized controlled trial will remotely enroll 60 subjects. Each participant will complete 20 stimulation sessions at a rate of 3-5 sessions per week. Each session will be 30 minutes on the day of usage. The study will be randomized with a 1:1 active; or sham control allocation. Endpoint analysis will be performed upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Report clinically significant symptoms of anxiety, defined as a score of 10 or greater on the Generalized Anxiety Disorder Scale, 7th edition (GAD-7)
* Males or females 18-80 years of age inclusive on starting the study
* Can speak/read English
* Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with trying to use the device on a daily basis
* Not using, and have never used, prescription, or the counter, anxiety medications
* Agree not to undergo any extreme lifestyle changes during the duration of the study that could impact sleep e.g. dietary or exercise changes

Exclusion Criteria:

* History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
* Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent the Modius Stress device from working)
* Medication for anxiety
* Use of beta-blockers within 1 month of starting the study
* Use of antidepressants or unstable dose within 3 months of starting study
* Use of any other medical condition or medication use that in the opinion of the PI is likely to make the participant resistant to VeNS.
* A score higher than 14 on the Insomnia Severity Index (ISI)
* A history of stroke or severe head injury (as defined by a head injury that required a craniotomy or endotracheal intubation). (In case this damaged the neurological pathways involved in vestibular stimulation).
* Presence of permanently implanted battery-powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator, etc.).
* Pregnancy or breast-feeding or intends to become pregnant (a pregnancy kit can be mailed if any uncertainty)
* History of epilepsy
* History of active migraines with aura
* History of head injury requiring intensive care or neurosurgery
* History of diagnosed cognitive impairment such as Alzheimer's disease/dementia
* History of bipolar, psychotic or substance use disorders
* Diagnosis of a current psychotic disorder
* Regular use (more than twice a month) of antihistamine medication within the last 6 months.
* History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas)
* A diagnosis of myelofibrosis or myelodysplastic syndrome.
* Previous use of any VeNS device
* Participation in other clinical trials
* History of vestibular dysfunction or another inner ear disease

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Generalised Anxiety Disorder (GAD-7) Scores | Up to 6 weeks
  To evaluate the ability of the Modius Stress device, relative to the control group, in the management of anxiety.

SECONDARY OUTCOMES:
Number of adverse events | Up to 6 weeks
  To evaluate the safety of the VeNS device relative to control group, in terms of the occurrence of adverse events.
Quality of life using SF-36 scores | Up to 6 weeks
Insomnia Severity Index (ISI) score | Up to 6 weeks
  To evaluate the effect of the VeNS device, relative to control group on participants with insomnia. ISI is a self-report rating scale assessing the severity of insomnia symptoms (range 0-28) with higher scores indicating a more severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Sailesh Kumar Goothy, Principal Investigator — R.D. Gardi Medical College, Ujjain, Madhya Pradesh.
Locations (1):
- Department of Psychiatry of R.D. Gardi Medical College, Ujjain, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No